CLINICAL TRIAL: NCT06531551
Title: "The Effect of Acupressure on Anxiety, Pain and Vital Signs in Gynecological Cancer Patients Receiving Brachytherapy: A Randomized Controlled Study"
Brief Title: The Effect of Acupressure on Patients Receiving Brachytherapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ülkü Saygılı, Assist. Prof, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18.04.24
Record Dates: First submitted 2024-04-18; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Brachytherapy; Complementary Approaches; Gynecological Cancers
Keywords: Brachytherapy; Acupressure; Nursing intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): Acupressure
  Interventions: Other: The group to which Acupressure will be applied in each fraction
- Control (No Intervention): Only routine practices of the clinic will be carried out

INTERVENTIONS:
Other: The group to which Acupressure will be applied in each fraction — Acupressure application protocol will be started after patient information. This process is planned to take 30 minutes.Before the application, approximately 20 seconds of warming and rubbing without direct pressure on the acupressure points will be performed to reduce tissue sensitivity and prepare the points for acupressure. Subsequently, the researcher will apply pressure with the thumb on the predetermined acupressure points, considering the individual's pain threshold, with 10 seconds of pressure followed by two seconds of relaxation without lifting the finger, in consecutive presses following the rhythm of breathing. A digital clock (belonging to the researcher) will be used to determine the duration of the acupressure application.
  Arms: Study

SUMMARY:
This study aimed to use acupressure to reduce anxiety in gynecologic cancer patients receiving brachytherapy. It was also aimed to investigate the effects of acupressure on anxiety, pain, and vital signs.

DETAILED DESCRIPTION:
Brachytherapy is a type of radiotherapy used in cancer treatment. In this method, the radiation source is placed directly on the tumor or the area to be treated. In this way, high doses of radiation are applied only to the target area, while surrounding healthy tissues are less damaged. Brachytherapy is usually used in the treatment of certain types of cancer, such as prostate, cervix, breast, and skin cancer. Gynecological brachytherapy is the application of brachytherapy in the treatment of gynecological cancers. It can be used especially in cancers of the uterus, cervix, vagina, and vulva. This treatment method is performed by placing the radiation source in the area where the tumor is located. Brachytherapy can be used in combination with surgery, chemotherapy, or other types of radiotherapy in the treatment of these types of cancers. Factors such as cancer burden, the problem of achieving remission, and the need for patients to remain immobile during the procedure, which is performed in a room that needs to be isolated due to radiation, contribute to symptoms such as pain and anxiety before and during treatment. These symptoms can sometimes affect vital signs. The need for patients to remain immobile during brachytherapy, the need to be isolated in a room due to radiation, and the discomfort caused by the applicators also increase anxiety in women. Patients often experience fear and anxiety because there is insufficient information about brachytherapy that could help relieve their pain and anxiety. Despite the complexity of such a procedure and the significant patient population, there are few studies on women's experiences with brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* Being registered in Selçuk University Faculty of Medicine Hospital Radiation Oncology Polyclinic
* Brachytherapy (intracavital brachytherapy) treatment protocol will be applied due to gynecological cancer.

to be

* Karnofsky Performance Scale being 80 and above (Performance scale for cancer patients)
* Being between the ages of 18 and 65
* Being conscious and cooperative
* Verbal and written approval to participate in the study after an explanation about the study is made.

Exclusion Criteria:

Impaired skin integrity in the acupressure application area

* Refuses to participate in the study after making a statement about the study.
* Bone or spine metastasis
* Amputation of the extremities to be applied
* Not having any mental illness

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory | day 1
  The Turkish validity and reliability of the State Anxiety Scale developed by Spielberger and his team in 1970 were conducted by Öner and Le Compte (1983). This scale is used to evaluate the emotional state that an individual feels at a specific moment and under specific conditions. The scale consists of 20 items and is evaluated on a four-point Likert scale (1-not at all, 2-somewhat, 3-very much, 4-completely). The scale includes both direct statements (3, 4, 6, 7, 9, 12, 13, 14, 17, 18) and reversed statements (1, 2, 5, 8, 10, 11, 15, 16, 19, 20).In direct statements, a value of 4 indicates high anxiety, while in reverse statements, a value of 1 signifies high anxiety. The total score range is 20-80, and this scoring is interpreted as follows: "no anxiety" between 0-19, "mild anxiety" between 20-39, "moderate anxiety" between 40-59, "severe anxiety" between 60-79, and a score of 80 is considered a "panic value.
Visual Analog Scale | day 1
  On a 10 cm ruler with "no pain" marked at one end and "worst pain imaginable" at the other, the patient indicates their perceived level of pain. The Visual Analog Scale (VAS) is reported to be more sensitive and reliable in assessing pain intensity compared to other single-dimensional scales in the measurement of pain severity according to the Numeric Rating Scale.
The Hospital Anxiety and Depression Scale | day 1
  The Hospital Anxiety and Depression Scale was developed by Zigmond and Snaith in 1983 (Zigmond AS & Snaith RP, 1983). It is stated that the scale is a reliable tool for detecting depression and anxiety in outpatient settings and provides valid measurements of the severity of emotional disorders through depression and anxiety subscales. In the scale consisting of 14 items, odd-numbered items investigate the anxiety sub-dimension, even-numbered items investigate the depression sub-dimension. It has a four-point Liket type feature between 0 and 3 points. Scoring for odd-numbered items 1, 3, 5, 6, 8, 10, 11 and 13 is 3, 2, 1, 0. Even items 2, 4, 7, 9, 12 and 14 are scored as 0,1,2,3. The scale score range is between 0-42. The cut-off score for the anxiety subscale was reported as 10, and the cut-off score for the depression subscale was reported as 7. Individuals who score above these scores constitute the risk group.
Vital signs | day 1
  Body temperature, Blood pressure, Pulse, Respiration; will be manually assessed by the researcher for 1 minute. Record will be made on the Personal Information Form.

CONTACTS AND LOCATIONS:
Overall Officials: ülkü Saygili Düzova, Study Director — Selçuk Üniversitesi Hemşirelik Fakültesi
Locations (1):
- ülkü Saygili Düzova, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duzova US, Can G, Duzova M, Basaran H, Yavas C. The effect of acupressure on anxiety, depression, pain, and vital signs in gynecological cancer patients receiving brachytherapy: A randomized controlled study. Support Care Cancer. 2025 Jul 18;33(8):698. doi: 10.1007/s00520-025-09754-6. PMID 40679634